CLINICAL TRIAL: NCT06658678
Title: Achieving Linkage to Retention and Treatment After Territory-wide Screening and Care Referral for Chronic Hepatitis B Patients
Brief Title: Linkage to Care and Treatment of Chronic HBV Patients
Acronym: HBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wai-Kay Seto, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HBVcare
Record Dates: First submitted 2024-06-25; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receiving an educational intervention (Experimental): Receiving the educational video link on their mobile device
  Interventions: Other: Receiving an educational intervention
- No educational intervention (No Intervention)

INTERVENTIONS:
Other: Receiving an educational intervention — Patient not receiving any educational intervention
  Other Names: No educational intervention
  Arms: Receiving an educational intervention

SUMMARY:
Chronic hepatitis B remains the leading cause of liver related mortality and morbidity globally and locally. Countries have been formulating initiatives to meet the WHO target of eliminating viral hepatitis by 2030. However, data on the most important aspect of management of chronic hepatitis B, namely linkage to care and treatment, remains scarce. In order to achieve the WHO goal, treatment rate of eligible patients should reach 80%.

DETAILED DESCRIPTION:
Diagnosing patients with chronic hepatitis B virus (HBV) infection and establishing linkage to treatment is important in achieving the World Health Organization (WHO) objectives in eliminating HBV as a public health threat by 2030. Global HBV diagnosis rates and treatment rates among eligible patients were 10% and 5% respectively. In Mainland China and Hong Kong, estimated diagnosis and treatment coverage were 19-27% and 11-22% respectively, similarly much lower than the WHO 2030 goals of 90% for diagnosis and 80% for treatment. A recent modeling study demonstrated that even if a modest 50% diagnosis rate was achieved in China, this will result in a 19% mortality decline, with 2.1 million deaths averted. Currently, HBV screening is recommended for persons born in regions with a HBV prevalence of 22%. This includes the vast majority of East Asian countries.

In the HBV care continuum, identifying patients and arranging linkage to care is only the first step. Long-term retention of patients is critical, especially since with disease progression, treatment eligibility rates can increase by 30% after 3 years of follow-up. Nonetheless, there has been a paucity of data on HBV care continuum retention rates after referrai and linkage. A US-based study did found that among diagnosed patients, only 63.2% achieved linkage to referral, and only 44.1% remained retained in clinical care after at least three clinic visits. Another study in Italy found a higher retention of 60% after 5 years; besides African ethnicity and concomitant HIV infection, the study failed to identify any predictors of retention failure, yet 74.8% of retained patients subsequently required treatment. There has been otherwise no published data on linkage to retention rates in endemic regions including East Asia, and on whether the care continuum cascade can successfully link referral to treatment.

Our center previously conducted a territory-wide prevalence study of HBV, and out of >10,000 screened participants, the investigators identified 803 hepatitis B surface antigen (HBSAg)-positive individuals, with a mean age of 53.7 (135.8) years (36.7% male). As part of linkage to care, all patients were subsequently referred to their respective geographical cluster hospital. The investigators recently performed a follow-up telephone survey of the 803 patients, asking on their status of clinical follow-up and liver-related treatment. Our preliminary data found a retention rate of only 37.1% after 2 years post-referral. However, among retained patients, 51.2% were already started on anti-HBV treatment, suggesting that high rates of treatment eligibility may also exist in unretained patients. Hence, to enhance linkage to treatment, linkage to retention rates will need improvement.

There is emerging evidence on the effect of different interventions in improving the care continuum of viral hepatitis, although the majority of evidence is concentrated in hepatitis C virus and not HBV. Clinical reminders have been demonstrated to be the most effective method to improve testing rates; such reminders may also be useful to in improving clinic attendance and retention. On the other hand, the data on educational materials is less consistent. Data was concentrated in Asian migrants in North America, with some based on non-randomized studies, and could be susceptible to selection, attrition and reporting bias.

Interventions using social media and mobile technology may be promising. Experience from engaging patients with human immunodeficiency virus infection have found social media effective in reaching out to marginalized individuals, especially among those of a younger age. It would be interesting to see if educational videos disseminated on mobile devices via social media can improve linkage to retention and treatment for HBV.

ELIGIBILITY:
Inclusion Criteria:

* CHB (HBV DNA+ or HBsAg+ for more than 6 months)
* Age >18
* Treatment naive at initial presentation

Exclusion Criteria:

* Prior HBV treatment
* Organ transplant or other immunosuppression
* HIV, HDV, HCV co-infection
* Decompensated or HCC patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The effect of education intervention on rate of retention in care in chronic hepatitis B patients identified from a territory wide screening program | 12 months

SECONDARY OUTCOMES:
The treatment rate in chronic hepatitis B patients up to 5 years after diagnosis | 5 years
The rate of viral suppression in chronic hepatitis B patients up to 5 years after diagnosis | 5 years
The rate of complication in chronic hepatitis B patients up to 5 years after diagnosis | 5 years
Factors affecting rate of retention in care from patient perspective in the form of questionnaire survey | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Department of Surgery, The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No